CLINICAL TRIAL: NCT01477658
Title: Effects of Chronic Right Ventricular Pacing in Children With Advanced Atrioventricular Block
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Roberto Costa, Associated Professor of Cardiovascular Surgery, University of Sao Paulo
Other Study IDs: CAPPesq nº 1248/09
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-05

CONDITIONS: Congenital Complete Atrioventricular Heart Block; High Grade Atrioventricular Block; Postoperative Complete Heart Block
Keywords: Congenital Complete Atrioventricular Heart Block; Pacemaker; Cardiac pacing; Children; Heart failure; Ventricular dyssynchrony; Echocardiography; Quality of life; Six-minute walk test; Young adults
MeSH Terms: conditions — Congenital heart block; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Congenital AV Block: Patients diagnosed with Congenital Complete Atrioventricular Heart Block
- Postoperative AV Block: Patients diagnosed with postoperative AV block

SUMMARY:
Recent studies have shown that chronic stimulation of the right ventricle can cause deleterious effects to cardiac function and synchronicity. The occurrence and consequences of this phenomenon in children and young patients with cardiac pacemaker due to advanced atrioventricular block (AVB) are still unknown.

Thus, our aims is to assess the chronic effects of cardiac pacing in children and young patients with advanced AVB and its impact on clinical, functional and echocardiographic parameters.

DETAILED DESCRIPTION:
This is a prospective cohort study that will include patients younger than 18 years-old at initial pacemaker implantation due to advanced AVB.

The design of the study will involve the following stages:

1. Screening and enrollment: patients will be selected consecutively during ambulatory care at our Institution or by the database of the Surgical Unity of Cardiac Pacing;
2. Clinical and laboratory evaluation: patient history, clinical evaluation, serum levels of neurohormonal and inflammatory biomarkers of heart failure, clinical and laboratory investigation of autoimmune rheumatic diseases, quality of life (SF-36, CHQ-PF50) and six-minute walk test;
3. Evaluation of ventricular function and cardiac synchronicity: Tissue Doppler (TDI) and real-time three-dimensional echocardiography (RT3DE);
4. Follow-up: patients will be monitored during 24 months.

The main end-points are:

* Clinical and functional changes (NYHA functional class)
* Heart failure hospitalization
* Quality of life
* Overall and cardiac mortality
* Cardiac resynchronization therapy and heart transplantation

ELIGIBILITY:
Inclusion Criteria:

* Age <18 years at initial pacemaker implantation
* Advanced AV block with /without congenital heart defects
* Time under cardiac pacing superior than one year
* Unicameral or atrioventricular pacing in single right ventricle site
* Informed consent of the patient or responsible

Exclusion Criteria:

* Bifocal or biventricular pacing
* Discontinuing use of the device for recovery of atrioventricular conduction
* Cardiac transplantation
* Inability to participate in the study procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ambulatory Care
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2007-11; Primary Completion 2012-11 (Actual); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Mortality | 24 months after enrollment

SECONDARY OUTCOMES:
Echocardiogram and Clinical Composite | baseline and 24 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Costa, MD, PhD, Study Chair — University of Sao Paulo; Roberto M Oliveira Jr, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Heart Institute (InCor) of University of São Paulo Medical School (Brazil), São Paulo, São Paulo, Brazil